CLINICAL TRIAL: NCT05151783
Title: Effects of Scapular Proprioceptive Neuromuscular Facilitation Techniques in Addition to Routine Physical Therapy on Clinical Outcomes in Patients With Adhesive Capsulitis:a Randomized Controlled Trial
Brief Title: PNF Technique in Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Shazib Butt, Principal investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 818-II
Record Dates: First submitted 2021-11-04; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; scapular PNF technique; shoulder range of motion
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy (Active Comparator): routine physical therapy for adhesive capsulitis
  Interventions: Other: conventional physiotherapy
- PNF techniques (Experimental): PNF techniques along with conventional physiotherapy
  Interventions: Other: PNF technique

INTERVENTIONS:
Other: conventional physiotherapy — Control group receivewill routine physical therapy including modalities like ultrasound (3 MHz continuous type; duration 10 minutes), heat modalities (apply to the involved region of shoulder joint shoulder for 10 minutes), shoulder ROM exercises, capsular stretching, and joint mobilization 5 times per week for four weeks. Duration of session will be 40 minutes.
  All Maitland mobilization will be given in supine position. After giving glenohumeral (GH) joint distraction, GH caudal glide, GH dorsal glide, and GH ventral glide were given at a rate of 2-3/second oscillations for 1-2 minutes to patients. Grade I or II rhythmic oscillations will be applied in pain free movement.
  Arms: conventional physiotherapy
Other: PNF technique — Group will receive scapular PNF techniques with routine physical therapy explained above For PNF techniques, patients will be lying on unaffected shoulder. In this group, 20 repetitions of diagonal scapular Pattern (Anterior Elevation and Posterior Depression and Posterior Elevation and Anterior Depression) with 20 sec rest period will be given to patients. Preparatory instructions for the desired movement will be given to patients at the start of procedure. PNF facilitation techniques of RI (Rhythmic initiation) & repeated contractions will be used in all patterns
  Arms: PNF techniques

SUMMARY:
Adhesive capsulitis is painful movement restricted condition linked with pain, restricted range of motion and difficulty in performing daily life activities. Multiple treatment options are there for its treatment. However, role of peripheral neuromuscular facilitation in this regimen is still under consideration.

DETAILED DESCRIPTION:
Adhesive Capsulitis or peri-arthritis or Frozen Shoulder is self-limiting condition of unknown etiology that usually affects middle aged population of 40-70 years and rarely it occur secondary to rheumatoid arthritis, osteoarthritis, trauma or immobilization of shoulder joint. It is characterized by development of dense adhesions, capsular thickening and restrictions which limits active and passive shoulder range of motion (ROM) with scapular dyskinesia.The aim of the of the study is to investigate the effects of scapular proprioceptive neuromuscular techniques with routine physical therapy on pain, scapular dyskinesia, shoulder ranges of motion and functionality in patients with adhesive capsulitis. Proper functioning of upper extremities requires both motion and stability of scapula on thorax. Prolonged immobilization of shoulder joint leads to ankylosis of joint and scapular dyskinesia. This study will help with a positive effect by using a non-invasive, less painful, cost effective and time saving approach of scapular proprioceptive neuromuscular facilitation techniques among joint mobilization and other therapeutic approaches like intra articular injections and manipulation under anesthesia on alleviating pain, muscle strength, shoulder ranges of motion and early restoration of normal functioning of shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of stage II & III adhesive capsulitis
* Referred by orthopedic physician
* Duration of stage approximately 1 month
* Both male and female
* Age: 40-70 years

Exclusion Criteria:

* Recent history of trauma
* Dislocation or fractures of shoulder
* History of diabetes and hypertension
* Congenital shoulder deformity
* Previous surgery patients
* Patients with diagnosed cardiovascular disease
* Patients with malignancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | Baseline data will be collected and then at 2nd week and 4th week.
  pain measured by visual analogue scale where o represents no pain and 10 represents severe pain
change in shoulder Range of motion | Baseline data will be collected and then at 2nd week and 4th week.
  shoulder range of motion through goniometer
change in shoulder functional activities | Baseline data will be collected and then at 2nd week and 4th week.
  shoulder functional activities by simple shoulder function test
change in scapular mobility | Baseline data will be collected and then at 2nd week and 4th week.
  scapular mobility through lateral scapular slide test

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad sh butt, Principal Investigator — University of Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckert AJ, Plaumann M, Pehlke S, Beck C, Muhldorfer S, Weickert U, Laimer M, Pfeifer M, Stechemesser L, Holl R. Idiopathic Frozen Shoulder in Individuals with Diabetes: Association with Metabolic Control, Obesity, Antidiabetic Treatment and Demographic Characteristics in Adults with Type 1 or 2 Diabetes from the DPV Registry. Exp Clin Endocrinol Diabetes. 2022 Jul;130(7):468-474. doi: 10.1055/a-1543-8559. Epub 2021 Aug 23. PMID 34425597
- [Result] Pandey V, Madi S. Clinical Guidelines in the Management of Frozen Shoulder: An Update! Indian J Orthop. 2021 Feb 1;55(2):299-309. doi: 10.1007/s43465-021-00351-3. eCollection 2021 Apr. PMID 33912325
- [Result] Prasanna KJ, Rajeswari R and Sivakuma V. Effectiveness of scapular proprioceptive neuromuscular facilitation (pnf) techniques in adhesive capsulitis of the Shoulder Joint. J Physiother Res 2017; 1: 9.
- [Result] Ebadi S, Forogh B, Fallah E, Babaei Ghazani A. Does ultrasound therapy add to the effects of exercise and mobilization in frozen shoulder? A pilot randomized double-blind clinical trial. J Bodyw Mov Ther. 2017 Oct;21(4):781-787. doi: 10.1016/j.jbmt.2016.11.013. Epub 2016 Nov 27. PMID 29037627
- [Result] Mishra N, Mishra A and Charaniya P. Effect of scapular proprioceptive neuromuscular facilitation on pain and disability in patients with adhesive capsulitis. Int J Yoga 2019; 4: 995-1000.
- [Result] Balci NC, Yuruk ZO, Zeybek A, Gulsen M, Tekindal MA. Acute effect of scapular proprioceptive neuromuscular facilitation (PNF) techniques and classic exercises in adhesive capsulitis: a randomized controlled trial. J Phys Ther Sci. 2016 Apr;28(4):1219-27. doi: 10.1589/jpts.28.1219. Epub 2016 Apr 28. PMID 27190456